CLINICAL TRIAL: NCT04488757
Title: Neurobiological Mechanisms of Stress in Youth With Chronic Widespread Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sarah Nelson, Assistant Professor and Attending Psychologist, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00035303; 1K23AT010643-01A1 (NIH)
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Widespread Pain; Stress, Psychological; Stress, Physiological
Keywords: Chronic Widespread Pain; Pediatric Pain; Allostatic Load; fMRI; Mind-Body Interventions
MeSH Terms: conditions — Chronic Pain; Stress, Psychological | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: All participants will undergo fMRI and stress physiology measurement. Intervention outcomes will be compared across two groups: 1. pediatric chronic widespread pain and 2. age and gender matched healthy controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Other): All participants enrolled in the study will undergo baseline fMRI and baseline and follow-up (4-month post-baseline) assessment of stress physiology (i.e., allostatic load). Treatment as usual information will be gathered for all participants to assess observational intervention response.
  Interventions: Diagnostic Test: functional Magnetic Resonance Imaging (fMRI); Other: Allostatic Load Composite

INTERVENTIONS:
Diagnostic Test: functional Magnetic Resonance Imaging (fMRI) — Participants will undergo a one hour fMRI scan with pain-induction using heat-based QST protocol.
Other: Allostatic Load Composite — All participants will be asked to provide saliva samples to measure cortisol response over time and dehydroepiandrosterone (DHEA) in addition to physiological measurements such as blood pressure/pulse, height/weight, and waist-hip ratio. Measurements will be taken at baseline and 4-month follow-up.

SUMMARY:
Chronic widespread pain (CWP) is a common chronic pain condition in youth and often associated with significant pain-related and psychosocial impairment. Understanding the neurobiological mechanisms that may underlie pediatric chronic pain and pain-related impairment can inform future treatments to ameliorate patients' suffering, making it a critical area of empirical investigation.

DETAILED DESCRIPTION:
Pediatric chronic widespread pain (CWP) is a serious public health problem resulting in high levels of healthcare utilization and disability. Youth with CWP also frequently report exposure to adverse childhood experiences (ACEs; abuse/neglect, violent/conflictual home environment, etc.) and a significant subset continue to experience physical and psychosocial impairment long-term. Certain mind-body interventions such as mindfulness-based stress reduction (MBSR) or meditation may be particularly appropriate for youth with CWP as they have been shown to modulate stress-induced maladaptation of the HPA-axis, autonomic nervous system, cardiovascular system, and brain structure (e.g., hippocampus). However, it is currently unknown if these targets are affected in youth with CWP. Preliminary research indicates that allostatic load (AL), or "wear and tear" on the nervous system due to stress, may contribute to pain chronicity. Similarly, evidence suggests that the hippocampus, a brain structure that is among the most deleteriously affected by stress, plays a role in pain perception. However, no study to-date has examined AL and hippocampal functioning in relation to stress exposure in youth with CWP. Mind-body interventions such as MBSR or meditation are an important and safe therapy option for both pain and stress reduction in youth with CWP and may modulate the negative impact of ACEs, so there is a critical need to know if these mechanisms are engaged in this population. The current study utilizes multifactorial physiological and neuroimaging measurement techniques to enhance our understanding of the potential role of these mechanisms in pain-related impairment and responsiveness to mind-body interventions over time. The aims of this study are to better characterize AL, assessed via a multifactorial composite, and hippocampal functioning via fMRI in pediatric CWP as specific targets for mind-body interventions that can lead to treatment optimization and improved compliance.

ELIGIBILITY:
Chronic Widespread Pain (CWP) group:

Inclusion Criteria:

* Between ages 11-17 years
* Referred to the Boston Children's Hospital Pain Treatment Service for evaluation of a CWP condition with duration > 3 months
* Right-handed

Exclusion Criteria:

* Inability to speak sufficient English to complete questionnaires
* Severe cognitive impairment
* Prescription steroidal (interference with cortisol measures) or psychotropic medication
* Any other chronic pain diagnosis (e.g., migraines, abdominal pain, CRPS)
* fMRI contraindications (e.g., dental appliances)

Healthy Control (HC) group:

Inclusion Criteria:

* Between ages 11-17 years
* Right-handed

Exclusion Criteria:

* Inability to speak sufficient English to complete questionnaires
* Severe cognitive impairment
* Prescription steroidal (interference with cortisol measures) or psychotropic medication
* Any chronic pain diagnosis
* Presence of documented chronic (> 3 months) medical condition with an identifiable, organic cause (e.g., diabetes, cystic fibrosis)
* fMRI contraindications (e.g., dental appliances)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Hippocampal Functioning | baseline
  measured via fMRI
Change in Morning Cortisol | baseline and 4-month follow-up
  measured via 2 samples of saliva taken via passive drool over the course of two days. After analysis, morning cortisol will be dichotomously coded with participants receiving a "1" if they score over one standard deviation above the mean. Coding will them be combined to formulate an allostatic load risk ratio, with higher scores indicating greater risk for allostatic load.
Change in Dehydroepiandrosterone (DHEA) | baseline and 4-month follow-up
  measured via 2 samples of saliva taken via passive drool over the course of two days. After analysis, DHEA will be dichotomously coded with participants receiving a "1" if they score over one standard deviation above the mean. Coding will them be combined to formulate an allostatic load risk ratio, with higher scores indicating greater risk for allostatic load.
Change in Flattened Cortisol | baseline and 4-month follow-up
  measured via 10 samples of saliva taken via passive drool over the course of two days. After analysis, the presence of cortisol will be dichotomously coded with participants receiving a "1" if the change in cortisol levels across the day fell at or below one standard deviation below the mean. Coding will them be combined to formulate an allostatic load risk ratio, with higher scores indicating greater risk for allostatic load.
Change in Blood Pressure | baseline and 4-month follow-up
  measured via blood pressure cuff by trained nurse. Results will be coded to capture levels that fall in the "normal", "prehypertension" and "hypertension" range with individuals scoring in the latter two ranges receiving a coding of "1" to be included in the allostatic load risk composite measure. Scoring of blood pressure ranges will be done using ezbmi- calculates deviation from expected BP/BMI by age/gender.
Change in Body-Mass Index (BMI) | baseline and 4-month follow-up
  measured via height and weight (in cm and kg) by a trained nurse. Results will be coded to capture individuals that score in the "underweight", "normal", "overweight" and "obese" ranges with individuals falling in all categories but "normal" receiving a coding of "1" to be included in the allostatic load risk ratio. Scoring of BMI ranges will be done using ezbmi- calculates deviation from expected BP/BMI by age/gender.
Change in Waist-Hip Ratio (WHR) | baseline and 4-month follow-up
  measured via tape measure around the smallest part of the waist and the widest part of the hips by a trained research coordinator. Results (waist measurement/hip measurement) will be coded dichotomously with individuals scoring a "1" whose WHR falls greater than or equal to one standard deviation above the mean of the sample. This scoring will also be included in the larger allostatic load risk ratio.
Change in Heart Rate (HR) | baseline and 4-month follow-up
  measured via pulse taken by a trained nurse. Results will be coded dichotomously with individuals scoring a "1" whose HR falls greater than or equal to one standard deviation above the mean of the sample. This scoring will also be included in the larger allostatic load risk ratio.

SECONDARY OUTCOMES:
Change in Pain Intensity | baseline and 4-month follow-up
  measured via numeric rating scale (range: 0-10). Higher rating indicates more intense pain.
Change in Functional Disability | baseline and 4-month follow-up
  measured via self-report Functional Disability Inventory (range: 0-60). Higher rating indicates greater functional disability.
Change in Sleep | baseline and 4-month follow-up
  measured via Patient Reported Outcome Measurement Information System (PROMIS) sleep disturbance scale short-form (8a). Raw scores are converted to T-scores (range: 0-100). Higher rating indicates greater impairment in sleep.

OTHER OUTCOMES:
Change in Treatment Engagement | baseline and 4-month follow-up
  measured via participant self-report of treatment as usual (e.g., engagement in physical therapy, cognitive-behavioral therapy, acupuncture, etc.). Observational measure without metrics for risk or impairment.
Change in Adverse Childhood Experiences (ACEs) exposure | baseline and 4-month follow-up
  measured via Childhood Trust Events Scale (CTES). Items on this measure are coded dichotomously (0 = no; 1 = yes) and will be summed to provide a total metric of ACEs exposure (range: 0-26).
Change in Psychological Stress | baseline and 4-month follow-up
  measured via Patient Reported Outcome Measurement Information System (PROMIS) psychological stress scale short-form (8a). Raw scores are converted to T-scores (range: 0-100). Higher rating indicates greater amounts of psychological stress.
Change in Anxiety | baseline and 4-month follow-up
  measured via Patient Reported Outcome Measurement Information System (PROMIS) anxiety scale short-form (8a). Raw scores are converted to T-scores (range: 0-100). Higher rating indicates greater amounts of anxiety.
Change in Depression | baseline and 4-month follow-up
  measured via Patient Reported Outcome Measurement Information System (PROMIS) depression scale short-form (8a). Raw scores are converted to T-scores (range: 0-100). Higher rating indicates greater amounts of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Nelson, Principal Investigator — Boston Children's Hospital/Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Nelson and collaborators acknowledge their willingness to share data and materials with other eligible investigators through academically established means.
  Finalized data sets will be available to other researchers who seek to conduct further analysis on any and all variables of the study, in full compliance with HIPAA and institutional IRB oversight. Interested researchers would need the permission of the PI of this study (Nelson). Any data-sharing agreement would include the purpose of the secondary analyses and the credentials of the researchers, and will be in full HIPAA compliance, as the data will be de-identified. This data-sharing agreement will meet the NIH's policy for data sharing.
Supporting Information: Analytic Code
Time Frame: Data will be made available on a case-by-case basis.